Date: 16/08/2017

<u>Study Title</u>: An investigation into the feasibility of incorporating an exercise rehabilitation programme for people with intermittent claudication into an already established Cardiac Rehabilitation service

## **Data Analysis:**

## **Quantitative data:**

The outcome data will be tested to see if it is normally distributed or not. SPSS software will then be used to assess for any statistically significant differences between the groups. Within groups and between group differences in exercise capacity will be analysed using a factorial ANOVA to compare the difference in the levels of improvement between groups. Wilcoxon tests will be used to analyse the questionnaire data.

The CAD group will also be compared to the National Audit of Cardiac Rehabilitation (NACR) data to assess the impact on the CAD group performance against expected national levels. The effect sizes will be calculated using the Cohen's *d* so that the results can be compared to other studies.

## **Qualitative Data:**

The analysis will be influenced by Braun & Clarke's (2006) six phases of thematic analysis as described in Table 2.

| Phase | Description of the process |
|---|---|
| 1. Familiarizing yourself with your | Transcribing data (if necessary), reading and re-reading |
| data: | the data, noting down initial ideas. |
| 2. Generating initial codes: | Coding interesting features of the data in a systematic |
| | fashion across the entire data set, collating data relevant |
| | to each code. |
| 3. Searching for themes: | Collating codes into potential themes, gathering all data |
| | relevant to each potential theme. |

| 4. Reviewing themes: | Checking if the themes work in relation to the coded extracts (Level 1) and the entire data set (Level 2), |
|---|---|
| 5. Defining and naming themes: | generating a thematic 'map' of the analysis. Ongoing analysis to refine the specifics of each theme, and |
| 5. Defining and naming themes. | the overall story the analysis tells, generating clear definitions and names for each theme. |
| 6. Producing the report: | The final opportunity for analysis. Selection of vivid, compelling extract examples, final analysis of selected extracts, relating back of the analysis to the research question and literature, producing a scholarly report of the analysis. |

Table 1 This table outlines the steps taken in the thematic analysis of the focus group data. Taken from: Braun & Clarke, (2006) Using thematic analysis in psychology. Qualitative Research in Psychology. 3: pp77-101

The results of both the quantitative data analysis and the thematic analysis from the focus groups will then be used to draw conclusions about the effectiveness of the treatment options.